CLINICAL TRIAL: NCT00541541
Title: Acoustic Cardiographic Assessment of Heart Function and the Role of Phrenic Nerve Stimulation Following Open Heart Surgery
Brief Title: Acoustic Cardiographic Assessment of Heart Function and the Role of Phrenic Nerve Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luzerner Kantonsspital (Other)
Collaborators: Inovise Medical (Industry)
Responsible Party: Principal Investigator, Prof. Paul Erne, Prof. Paul Erne, Luzerner Kantonsspital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Audicor-Pacing
Record Dates: First submitted 2007-10-08; First posted 2007-10-10 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Heart Failure, Congestive; Cardiac Pacing, Artificial; Transcutaneous Electric Nerve Stimulation
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Phrenic nerve stimulation — Patients receive a phrenic nerve stimulation

SUMMARY:
In this study, the investigators sought to determine whether a stimulation of the phrenic nerve affects heart function. Heart function is assessed by acoustic cardiography.

DETAILED DESCRIPTION:
Patients who need temporary pacing following open heart surgery and who are willing to participate receive a phrenic nerve electrode during the operation. Heart function is postoperatively assessed by acoustic cardiography (Audicor, Inovise Medical Inc., Portland, USA) during different forms of pacing (right ventricle, left ventricle, biventricular; AAI, DDD) and with or without phrenic nerve stimulation. Acoustic cardiography simultaneously integrates heart sounds and single-channel electrocardiography input to generate multiple parameters that correlate to established hemodynamic measures. Effects of phrenic nerve stimulation on heart function will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients following open heart surgery who need temporary pacing

Exclusion Criteria:

* Patients with permanent pacemakers
* Patients with fast changing need of vasopressor therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-02; Primary Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Change of electrical mechanical activation time (EMAT) as measure of heart function on different settings of pacing | One day

CONTACTS AND LOCATIONS:
Overall Officials: Paul Erne, MD, Study Chair — Luzerner Kantonsspital
Locations (1):
- Kantonsspital Luzern, Department of Cardiology, Lucerne, Canton of Lucerne, Switzerland